CLINICAL TRIAL: NCT02471053
Title: Exercise to Prevent AnthrCycline-based Cardio-Toxicity Study (EXACT)
Brief Title: Exercise to Prevent AnthrCycline-based Cardio-Toxicity Study
Acronym: EXACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Scott Grandy, PhD, Assistant Professor, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXACT2015
Record Dates: First submitted 2015-05-11; First posted 2015-06-12 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Neoplasms; Heart; Disease, Functional; Inflammation
Keywords: Exercise; Quality of Life; Complementary Therapies; Neoadjuvant Therapy; Feasibility Studies
MeSH Terms: conditions — Neoplasms; Disease; Inflammation; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Moderate Intensity Exercise (Experimental): All consenting patients will participate in an aerobic training program, twice-weekly over a 12-week period. Assessments will be performed at baseline (pre-training) and post-program (12-weeks). All participants will continue to receive standard care for their cancer diagnosis.
  Interventions: Other: Moderate Intensity Exercise

INTERVENTIONS:
Other: Moderate Intensity Exercise — Exercise sessions will be held twice-weekly and will begin with a group warm-up activity, followed by 45 minutes of aerobic activity and ending with a cool down. All aerobic exercise will be performed at a moderate intensity, defined as exercise that elicits a heart rate (HR) between 40-60% of heart rate reserve (HRR). Prior to the initial exercise session target heart rates will be calculated for each subject based on the maximum HR achieved during their baseline stress test.

SUMMARY:
As the numbers of cancer survivors grow, the long-term adverse effects of cancer therapy are becoming increasingly apparent. Most prominent are the toxic effects on the heart (cardiotoxicity) which may lead to cardiac dysfunction and increased risk of cardiovascular disease (CVD). The investigators hypothesize that an individualized aerobic training program for cancer patients receiving active treatment will be both feasible and safe and will result in improvements in overall levels of physical activity and quality of life.

Feasibility will be assessed by evaluating the recruitment, adherence and attrition rates, along with program safety. Efficacy will be assessed by evaluating changes in health-related outcomes.

DETAILED DESCRIPTION:
As the numbers of cancer survivors grow, the long-term adverse effects of cancer therapy are becoming increasingly apparent. Most prominent are the toxic effects on the heart (cardiotoxicity) which may lead to cardiac dysfunction and increased risk of cardiovascular disease (CVD). Of note, data indicate that the magnitude of CVD risk for long-term survivors may exceed the risk of a secondary malignancy, which is a known complication of primary cancer therapy. While long-term follow-up data in adult cancer survivors is lacking, study of adult survivors of childhood cancers shows that these individuals are 15 times more likely to develop congestive heart failure (CHF), 10 times more likely to develop CVD, and 9 times more likely to suffer a stroke compared individuals who have not had cancer. Thus, it is clear that the long-term cardiotoxic effects of cancer therapy represent a significant concern for cancer survivors. The mechanisms responsible for the damaging effects of cancer therapy are not fully understood, however there is a need to maximize the benefits of treatment while minimizing long-term damage. Recent animal studies suggest that aerobic exercise training may offer a protective effect against chemotherapy-induced heart disease. However, to the investigator's knowledge, no study to date has examined the potential cardioprotective benefits of exercise training for patients receiving cancer treatment.

Accordingly, the purpose of this pilot study is to evaluate the feasibility and efficacy of a 12-week supervised exercise program based on the principles of cardiac rehabilitation for patients receiving anthracycline-based chemotherapy.

Feasibility will be assessed by evaluating three outcomes, recruitment rate, adherence rate (i.e. exercise class attendance records), attrition rate, and safety (i.e. number of adverse events).

Efficacy will be assessed by evaluating changes in health-related outcomes to assess if these changes are equal to or better than what was measured at baseline. The health-related outcomes include cardiac function and biological markers of cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria - Only those patients who meet the following inclusion will be asked to participate in the study:

* Between the ages of 18 and 65;
* Receiving anthracycline chemotherapeutic treatment for a primary/non-recurrent breast or hematological malignancy;
* Are scheduled to received a minimum dose of 100 mg/m2 of doxorubicin (DOX) or 120 mg/m2 of daunorubicin (DAUN), or 150 mg/m2 epirubicin (EPI)
* Within eight weeks of first anthracycline dose;
* Do not have a previous history of myocardial infarction, cerebrovascular disease, peripheral vascular disease, congestive heart failure, or cardiomyopathy (controlled hypertension is not exclusionary);
* Have no known contraindications to light-to-moderate exercise;
* Have no known contraindications to cardiopulmonary exercise stress testing;
* Able to participate in the 12-week community-based exercise program;
* Provided medical consent from their treating physician

Exclusion Criteria:

* Any patients who meet the inclusion criteria, but have any significant cognitive limitations will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by rate of recruitment | 12 Weeks
  The rate of recruitment will be measured by comparing the number of patients screened to the number of patients enrolled (patients per month).
Number of adverse events | 12 Weeks
  The number of adverse events associated with exercise program will be used to examine safety.

SECONDARY OUTCOMES:
Feasibility as measured by program adherence | 12 Weeks
  The program adherence will be calculated by dividing the total number of exercise sessions by the number of actual session attended.
Feasibility as measured by attrition rate | 12 Weeks
  The attrition rate will be measured by the number of patients who drop out of the study.
Cardiac Function | 12 Weeks
  Cardiac function will be measured by examining heart chamber size, ventricular function and blood flow between the cardiac chambers using a Multigated acquisition (MUGA) scan.
Cardiac Disease Risk | 12 Weeks
  Cardiac disease risk will be measured using the Framingham Risk Score.
Aerobic Fitness | 12 Weeks
  Aerobic fitness will be measured by comparing baseline and 12 week cardiac stress tests and the associated peak oxygen uptake values.
Fatigue | 12 Weeks
  The Functional Assessment of Cancer Therapy - Fatigue questionnaire will be used to compare baseline and 12 week self-reported levels of fatigue.
Physical Activity Behaviours | 12 Weeks
  Baseline and 12 week levels of physical activity will be measured using the International Physical Activity Questionnaire.
Life Quality | 12 Weeks
  The Functional Assessment of Cancer Therapy - General questionnaire along with the appropriate tumor specific appendix, will be used to compare baseline and 12 week quality of life measures.
Lipid Profile | 12 Weeks
  Baseline and 12 week levels will be compared.
Fasting Glucose | 12 Weeks
  Baseline and 12 week levels will be compared.
High-sensitivity Troponin (hs-TNT) | 12 Weeks
  Baseline and 12 week levels will be compared.
N-terminal of the prohormone brain natriuretic peptide (NTproBNP) | 12 Weeks
  Baseline and 12 week levels will be compared.
C-reactive protein (CRP) | 12 Weeks
  Baseline and 12 week levels will be compared.
Cytokines (IL-1α) | 12 Weeks
  Baseline and 12 week levels (picogram per milileter) will be compared.
Cytokines (IL-1β) | 12 Weeks
  Baseline and 12 week levels (picogram per milileter) will be compared.
Cytokines (IL-4) | 12 Weeks
  Baseline and 12 week levels (picogram per milileter) will be compared.
Cytokines (IL-6) | 12 Weeks
  Baseline and 12 week levels (picogram per milileter) will be compared.
Cytokines (IL-10) | 12 Weeks
  Baseline and 12 week levels (picogram per milileter) will be compared.
Cytokines (IL-17) | 12 Weeks
  Baseline and 12 week levels (picogram per milileter) will be compared.
Cytokines (TNFα) | 12 Weeks
  Baseline and 12 week levels (picogram per milileter) will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Grandy, PhD, Principal Investigator — Assistant Professor, Affiliate Scientist, Division of Cardiology, Nova Scotia Health Authority
Locations (1):
- QEII Health Science Center, Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albini A, Pennesi G, Donatelli F, Cammarota R, De Flora S, Noonan DM. Cardiotoxicity of anticancer drugs: the need for cardio-oncology and cardio-oncological prevention. J Natl Cancer Inst. 2010 Jan 6;102(1):14-25. doi: 10.1093/jnci/djp440. Epub 2009 Dec 10. PMID 20007921
- [Background] Yeh ET. Cardiotoxicity induced by chemotherapy and antibody therapy. Annu Rev Med. 2006;57:485-98. doi: 10.1146/annurev.med.57.121304.131240. PMID 16409162
- [Background] Oeffinger KC, Mertens AC, Sklar CA, Kawashima T, Hudson MM, Meadows AT, Friedman DL, Marina N, Hobbie W, Kadan-Lottick NS, Schwartz CL, Leisenring W, Robison LL; Childhood Cancer Survivor Study. Chronic health conditions in adult survivors of childhood cancer. N Engl J Med. 2006 Oct 12;355(15):1572-82. doi: 10.1056/NEJMsa060185. PMID 17035650
- [Derived] Keats MR, Grandy SA, Giacomantonio N, MacDonald D, Rajda M, Younis T. EXercise to prevent AnthrCycline-based Cardio-Toxicity (EXACT) in individuals with breast or hematological cancers: a feasibility study protocol. Pilot Feasibility Stud. 2016 Aug 5;2:44. doi: 10.1186/s40814-016-0084-9. eCollection 2016. PMID 27965861